CLINICAL TRIAL: NCT00007891
Title: Phase I Study of 90-Y-Humanized-BrE-3 Followed by Autologous Hematopoietic Progenitor Cell Support in Patients With Metastatic Breast Cancer
Brief Title: Radiolabeled Monoclonal Antibody Therapy Followed by Bone Marrow or Peripheral Stem Cell Transplantation in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research Institute of Contra Costa (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CRICC-BB-IND-7186; CDR0000068340 (Registry Identifier: PDQ (Physician Data Query)); UCHSC-97467; NCI-V00-1637
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2004-09

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Filgrastim; Peripheral Blood Stem Cell Transplantation; Indium

INTERVENTIONS:
Biological: filgrastim
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: indium In 111 monoclonal antibody BrE-3
Radiation: yttrium Y 90 monoclonal antibody BrE-3

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Peripheral stem cell transplantation or bone marrow transplantation may be able to replace immune cells that were destroyed by monoclonal antibody therapy used to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of radiolabeled monoclonal antibody therapy followed by bone marrow or peripheral stem cell transplantation in treating patients who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of yttrium Y 90 labeled, humanized monoclonal antibody BrE-3 when given in combination with indium In 111 labeled, humanized monoclonal antibody BrE-3 followed by autologous bone marrow or peripheral blood stem cell transplantation in patients with metastatic breast cancer.
* Determine hematopoietic engraftment in these patients treated with this regimen.
* Determine the ability of indium In 111 labeled, humanized monoclonal antibody BrE-3 to image metastatic disease in these patients.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine the preliminary antitumor response in these patients treated with this regimen.

OUTLINE: This is a dose escalation study of yttrium Y 90 labeled, humanized monoclonal antibody BrE-3 (Y90 huMOAB BrE-3).

Patients receive Y90 huMOAB BrE-3 and indium In 111 labeled, humanized monoclonal antibody BrE-3 IV over 1-2 hours on day -14. Patients undergo autologous bone marrow or peripheral blood stem cell transplantation on day 0. Patients also receive filgrastim (G-CSF) IV beginning on day 0 and continuing until blood counts recover.

Cohorts of 3-6 patients receive escalating doses of Y90 huMOAB BrE-3 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicities.

Patients are followed every 3-4 months for 1 year and then at least annually thereafter.

PROJECTED ACCRUAL: Approximately 3-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic breast cancer

  * BrE-3 positive
  * Relapsed or refractory disease with tumor progression after effective therapy allowed
* Measurable or evaluable disease
* Received at least one prior chemotherapy regimen for metastatic disease and have at least one of the following:

  * Chemotherapy refractory liver metastases more than 2 cm
  * Multiple non-resectable liver metastases
  * Brain metastases
  * Prior high-dose chemotherapy
  * Relapse within prior radiotherapy field
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Over 18

Sex:

* Male or female

Menopausal status:

* Not specified

Performance status:

* 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,000/mm3
* Absolute neutrophil count greater than 1,000/mm3
* Platelet count greater than 100,000/mm3

Hepatic:

* Bilirubin less than 2 times normal
* SGOT/SGPT less than 2 times normal

Renal:

* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* LVEF greater than 45% by MUGA scan

Pulmonary:

* DLCO and FEV 1.0 greater than 60% predicted

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known hypersensitivity to E. coli derived proteins
* No other comorbid condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior high-dose chemotherapy with autologous peripheral blood stem cell transplantation

Chemotherapy:

* See Disease Characteristics
* See Biologic therapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* Not specified

Other:

* Recovered from prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-06; Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto L. Ceriani, MD, PhD, Study Chair — Cancer Research Institute of Contra Costa
Locations (2):
- United States (2):
  - Cancer Research Institute of Contra Costa, San Francisco, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado